CLINICAL TRIAL: NCT06411535
Title: Impact of Ultra-Processed Food Intake on Gingival Tissue Health: A Pre-post Clinical Study
Brief Title: Impact of Ultra-Processed Food Intake on Gingival Tissue Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Associate Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UPF001
Record Dates: First submitted 2024-05-01; First posted 2024-05-13 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Gingivitis; Ultra-processed Food; Prevention
MeSH Terms: conditions — Gingivitis | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients answer the OHIP 14 and the Food Frequency Questionnaires, and are classified according to the NOVA classification. A full-mouth periodontal chart is performed.
  After 8 weeks, Questionnaires are re-administered. A full-mouth periodontal chart is performed, along with a session of full-mouth ultrasonic debridement.
  After 16 weeks from baseline, administration of the OHIP 14 and the FFQ is repeated. Clinical variables are re-evaluated.
  Interventions: Other: Full-mouth ultrasonic debridement
- Nutritional Counseling Group (Experimental): Patients answer the OHIP 14 and a Food Frequency Questionnaires, and are classified according to the NOVA classification. A full-mouth periodontal chart is perfomed. Patients receive a nutritional counseling on the significance of reducing ultra-processed food intake. Patients receive weekly motivational emails, as part of the dietary counseling.
  After 8 weeks, Questionnaires are readministered. A full-mouth periodontal chart is performed, along with a session of full-mouth ultrasonic debridement. Nutritional counseling is reinforced. Patients receive weekly motivational emails, as part of the dietary counseling.
  After 16 weeks from baseline, administration of the OHIP 14 and the FFQ is repeated. Clinical variables are re-evaluated.
  Interventions: Behavioral: Full-mouth ultrasonic debridement plus Nutritional counseling

INTERVENTIONS:
Behavioral: Full-mouth ultrasonic debridement plus Nutritional counseling — After diagnosis of gingivitis, patients will receive a nutritional counseling focused on ultra-processed foods entails educating individuals about the nutritional content and potential health implications of highly processed food products. They will undergo a session of full-mouth ultrasonic debridement and reinforcment of dietary counseling. Between consecutive time points, patients will receive motivational emails.
  Arms: Nutritional Counseling Group
Other: Full-mouth ultrasonic debridement — After diagnosis of gingivitis, patients will receive a session of full mouth ultrasonic debridement
  Arms: Control Group

SUMMARY:
The shift towards consuming more industrialized food products, particularly ultra-processed foods, has been linked to a rise in non-communicable diseases globally. These products are energy-dense, high in unhealthy components, and often lead to overconsumption due to their palatability and convenience. Studies suggest a connection between ultra-processed food consumption and various health issues, including obesity and cardiovascular diseases. The present study is designed as a single-center, double-blind, parallel-arm randomized clinical trial. This study aims to investigate the impact of ultra-processed food consumption on gingival health and to evaluate the potential benefits of dietary counseling and reduced ultra-processed food intake on gingival inflammation over a 4-month period.

DETAILED DESCRIPTION:
The impact of shifting of a diet from less industrialized food products toward a more industrialized food products has a positive relationship to the global burden of non- communicable disease. This increase in the consumption of Ultra-Process food was first started in the high-income countries and now in medium-income countries. All together, they are energy dense, high in unhealthy types of fat, refined starches, free sugars and salt, and poor sources of protein, dietary fibre. Ultra-processed products are made to be hyper-palatable and attractive, with long shelf-life and able to be consumed anywhere, any time. Their formulation, presentation and marketing often promote overconsumption. Due to the high levels of additives, sugars and preservatives, they have been associated with various non-communicable diseases, including obesity, cardiovascular diseases and systemic inflammation like periodontitis. In order to investigate a relationship between ultra-process food consumption and gingival health we used a food frequency questionnaire conducted and evaluated in a study in south of Italy with the classification of food according to the NOVA classification.

In recent years the effect of ultra-processed foods consumption on systemic and oral health has received more attention. Several studies have reported a significant association between caries and ultra-processed food. However, the effect of an highly processed food diet on gingival tissues health has not been fully investigated. Thus, the aim of the present study is to assess the impact of ultra-processed food consumption on gingival inflammation

Primary Objective:

To assess the association between ultra-processed food intake and the health of gingival tissues of a University-based cohort of individuals

Secondary Objectives:

To determine the role of dietary counselling and reduced ultra-processed food consumption on the resolution of gingival inflammation.

Trial design The current protocol is designed as single-centre, double-blind, parallel arm, University-based, superiority, clinical trial with a 4-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years of age.
* Non-smokers (never smokers or former smokers for at least 6 months).
* Presence of FMBS >= 10%
* No interproximal attachment loss of ≥3 mm in ≥2 non-adjacent teeth

Exclusion Criteria:

* Carious lesions and/or inadequate restorations.
* Subjects currently undergoing orthodontic therapy or wearing occlusal bite guards.
* Subjects suffering any systemic disease or condition which may affect the response of gingival tissues or the ability to perform adequate plaque control (pregnancy, diabetes, quantitative and/or qualitative polymorphonuclear neutrophils defects, other immune system disorders, etc.)
* Subjects taking medications that could interfere with the gingival tissues response (i.e. anti-inflammatory agents, diphenylhydantoin, calcium channel blockers, cyclosporin A, immunostimulants/immunomodulators)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Change in Full Mouth Bleeding Score (FMBS) | Full Mouth Bleeding Score (FMBS) collected six sites per tooth, full mouth, will be recorded by a calibrated and blinded examiner at the baseline visit (T0), at two months (T2) and follwing active treatment, at 4 months (T4)
  Evaluate the effect of Nutritional Counseling on gingival bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Discepoli, DDS MSc PhD, Principal Investigator — Department of Medical Biotechnologies, University of Siena
Locations (1):
- AOUS, Siena, Italy